CLINICAL TRIAL: NCT03938740
Title: An Exploratory Randomized Open-Label 2-Arm Comparison of Insulin Dosing Algorithms Using Hepatic Directed Vesicle-Insulin Lispro and Insulin Degludec to Determine Optimum Basal Insulin Dosing Regimens in Type 1 Diabetes Mellitus Subjects
Brief Title: Comparison of Different Insulin Dosing Algorithms Using Hepatic Directed Vesicle-Insulin Lispro and Insulin Degludec
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Diasome Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DP 01-2019-01
Record Dates: First submitted 2019-04-15; First posted 2019-05-06 (Actual); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — insulin degludec

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- HDV-Insulin Lispro and Insulin Degludec dose reduced by 40% (Experimental): HDV-Insulin Lispro and Insulin Degludec dose reduced by 40%
  Interventions: Drug: HDV-Insulin Lispro and Insulin Degludec (-40%)
- HDV-Insulin Lispro and Insulin Degludec dose reduced by 10% (Experimental): HDV-Insulin Lispro and Insulin Degludec dose reduced by 10%
  Interventions: Drug: HDV-Insulin Lispro and Insulin Degludec (-10%)

INTERVENTIONS:
Drug: HDV-Insulin Lispro and Insulin Degludec (-40%) — HDV-Insulin Lispro and Insulin Degludec (-40%)
  Arms: HDV-Insulin Lispro and Insulin Degludec dose reduced by 40%
Drug: HDV-Insulin Lispro and Insulin Degludec (-10%) — HDV-Insulin Lispro and Insulin Degludec (-10%)
  Arms: HDV-Insulin Lispro and Insulin Degludec dose reduced by 10%

SUMMARY:
Multi-center, open-label, multiple dose safety, tolerability and efficacy study

DETAILED DESCRIPTION:
This is a 24-week, open-label, multiple dose safety, tolerability and efficacy study. There is a 12-week run-in phase when all subjects receive Insulin Lispro and Insulin Degludec for 12 weeks. After completing the run-in period, subjects then are randomized to a treatment group of either HDV- Insulin lispro + Insulin Degludec (Degludec dose reduced by 40%) or HDV-Insulin lispro+ Insulin Degludec (Degludec dose reduced by 10%) for 12 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female of age 18 to 65 years, inclusive.
2. If female of child-bearing potential, must agree for the duration of the study. to use adequate contraceptive measures, such as, intra-uterine device [IUD], oral or injectable contraceptives, or barrier method plus spermicide.
3. Has at Screening been diagnosed as T1DM for at least 12 months.
4. Has at Screening C-peptide ≤0.8 ng/mL (single retest allowed).
5. Has at Screening been on treatment with rapid analog insulin for the previous six (6) months.
6. Has at Screening willingness to use continuous glucose monitoring (CGM) technology throughout study.
7. Is, for the duration of the study, willing to use insulin lispro as the only analog bolus insulin and insulin degludec as the only basal insulin.
8. Has at Screening a BMI ≥18.0 kg/m2 and ≤33.0 kg/m2.
9. Has at Screening HbA1c ≥6.5% and ≤8.5%.

Exclusion Criteria:

1. Has known or suspected allergy to any component of any of the study drugs in this trial.
2. Is, at Screening, pregnant or breast-feeding, or intends to become pregnant at any time during the duration of the study.
3. Has, at Screening, as judged by the Site Investigator, a history or current evidence of any of the following complications of diabetes: proliferative retinopathy or maculopathy, severe neuropathy (in particular, autonomic neuropathy), symptomatic gastroparesis.
4. Is, at Screening, judged by the Site Investigator to have a current addiction to alcohol or substances of abuse.
5. Is, at Screening, using one or more drugs that may interfere with the interpretation of trial results or are known to cause clinically relevant interference with insulin action, glucose utilization, or recovery from hypoglycemia (e.g., beta blockers, systemic corticosteroids at pharmacologic doses, cancer chemotherapies.).
6. Has at Screening any of the following findings, unless approved by both the Site Investigator and the Medical Monitor:

   * Uncontrolled hypertension, defined as diastolic blood pressure ≥ 100 mmHg and/or systolic blood pressure ≥ 160 mmHg after 5 minutes in the sitting position;
   * History of or findings on EKG of cardiac arrhythmia or conduction defect;
   * Clinically significant abnormalities on Screening laboratory studies
7. Has, within one (1) month prior to Screening, used either oral anti-diabetic medication or non-insulin anti-diabetic injection therapies (e.g. SGLT-2 inhibitors, pramlintide, GLP-1 agonists, etc.).
8. Has, within one (1) month prior to Screening, received any investigational drug.
9. Has, within two (2) months prior to Screening, used an insulin pump delivery system.
10. Has, within three (3) months prior to Screening, smoked tobacco or used any smokeless tobacco or nicotine delivery system (inhaled, oral or buccal).
11. Has at Screening, as judged by the Site Investigator, any condition (intrinsic or extrinsic) that could reasonably be expected to interfere with trial participation, confound evaluation of the data, or pose additional risk to adhering to the study protocol. Examples of such conditions include but are not limited to:

    * Clinically significant active disease of the gastrointestinal, cardiovascular, hepatic, neurological, renal, genitourinary, or hematological systems;
    * History of such an illness or disease
    * Diminished mental capacity, psychological or behavioral dysfunction, unwilling or resistant to protocol requirements, language barriers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2019-03-18 (Actual); Primary Completion 2019-12-06 (Actual); Study Completion 2020-03-18 (Actual)

PRIMARY OUTCOMES:
Basal, bolus and total insulin doses (UOM=units) during the last 2 weeks of the treatment period | 24 weeks
  Basal, bolus and total insulin doses (UOM=units) during the last 2 weeks of the treatment period
Basal/bolus ratios during the last 2 weeks of the treatment period | 24 weeks
  Basal/bolus ratios during the last 2 weeks of the treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Marc Penn, MD, PhD, Study Director — Diasome Pharmaceuticals
Locations (7):
- United States (7):
  - Mills-Peninsula Medical Center, Diabetes Research Institute, San Mateo, California
  - Barbara Davis Center for Diabetes, Aurora, Colorado
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Endocrine Research Solutions, Inc., Roswell, Georgia
  - Diabetes & Endocrinology Consultants, PC, Morehead City, North Carolina
  - Texas Diabetes & Endocrinology, PA, Austin, Texas
  - Texas Diabetes & Endocrinology, PA, Round Rock, Texas

IPD SHARING:
Plan to Share IPD: No